CLINICAL TRIAL: NCT01012518
Title: Video-guided Percutaneous Tracheostomy (PCT): Evaluating the Safety, Efficacy and Simplicity of a Novel Technique, Compared to Conventional PCT
Brief Title: Video-guided Percutaneous Tracheostomy (PCT) Versus Conventional PCT: Comparing Safety and Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Patrick Sorkine, Intensive Care unit, Tel aviv Sourasky Medical center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TASMC-09-PS-0544-CTIL
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Bleeding; Hypoxia; Atelectasis; Pneumothorax; Pneumomediastinum
Keywords: percutaneous tracheostomy; paratracheal insertion; tracheal injury; transtracheal needle; ventilatory parameters
MeSH Terms: conditions — Hemorrhage; Hypoxia; Pulmonary Atelectasis; Pneumothorax; Mediastinal Emphysema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional PCT (Active Comparator): PCT performed without video guidance, as conventionally performed
  Interventions: Device: Standard PCT
- Video-assisted PCT (Experimental): PCT performed with the guidance of a camera-embedded ETT wired to a monitor
  Interventions: Device: Video-guided PCT

INTERVENTIONS:
Device: Standard PCT — The standard technique, performed without video guidance
  Other Names: Control; Conventional PCT
  Arms: Conventional PCT
Device: Video-guided PCT — PCT performed with the guidance of a camera-embedded ETT wired to a monitor
  Other Names: Video-assisted PCT; ETView-guided PCT
  Arms: Video-assisted PCT

SUMMARY:
The purpose of this study is to compare the feasibility, safety, efficacy and ease of performance of a video-assisted PCT (via an endotracheal tube embedded with a mini video-camera) with the standard ("blind") PCT technique.

DETAILED DESCRIPTION:
Background

Percutaneous tracheostomy (PCT) is commonly used in critically-ill patients who require long-term mechanical ventilation in the intensive care unit (ICU). While being effective and safe, this technique has some complications. These include paratracheal insertion of the tracheostomy tube, tracheal injury; puncturing the cuff and transfixing the endotracheal tube (ETT) during the transtracheal needle insertion; inserting the guide wire through Murphy's eye; or accidental extubation while withdrawing the endotracheal tube during the procedure leading to loss of the airway [1-6].

Although using the fingertip to palpate the trachea and endotracheal tube is a useful technique to locate the tip of the endotracheal tube during the procedure, it is unreliable, particularly in patients with short and thick necks. There are reports of lower rates of acute complications under endoscopic (bronchoscopic) guidance [7-11]. However, there is no adequate controlled study showing that endoscopic-guided tracheostomy is superior to the 'blind' one. Moreover, it is an expensive tool which is not readily available in some centers.

Video guidance provides a cost-effective alternative to bronchoscopes, that may also reduce the risk of procedure-related complications such as paratracheal insertion of the tracheostomy tube, tracheal injury or cuff puncture [12].

The goal of this study is to evaluate the safety, efficacy and operability of video-guided PCT compared with standard PCT. Video-guided PCT, a bedside safe and simple technique that can be performed in the ICU without the assistance of a pulmonologist, may overcome some of the limitations of the standard percutaneous tracheostomy.

The technique is based on the ETView TVTTM, a commercially available ETT, embedded with a mini video-camera at the tip of the tube. It provides direct endoscopic visualization of the larynx and tracheal mucosa, and thereafter allows the determination of the tip of the transtracheal needle during percutaneous puncture of the trachea, and hence may reduce the likelihood of paratracheal insertion, tracheal injury, or other technical complications.

The ETView TVTTM device is compatible with any medical grade NTSC video monitor, thereby it provides monitoring of the airways during the intubation and PCT procedure, as well as continuous viewing of the airways as long as mechanical ventilation is required.

Study Objectives To compare video-guided PCT to the standard technique in terms of success rate, efficacy, safety, and outcomes..

Study design The study will be conducted as a comparative, semi-blinded, matched one (according to sex, age and difficult airway - that will be assessed according to neck diameter and anatomical parameters). The setting will be the ICU of the Sourasky medical center. 60 consecutive adult critically ill patients who require elective tracheostomy will be recruited for the study. Informed consent will be obtained from the families or next of kin of all study patients. In the absence of relatives, consent will be given by an anesthesiologist/intensivist not related to the study. Both procedures will be performed by the same team of intensivists upon all study patients. During and following the procedure we will assess all of the parameters mentioned above.

Methods

The procedure

The procedure will be performed by an ICU team which includes: an anesthesiologist/intensivist who executes the procedure, another anesthesiologist who applies anesthetics & analgesia, a nurse, and a forth person who takes time.

During the procedures (either standard PCT or video-guided PCT) oxygen saturation, end tidal carbon dioxide (ETCO2), ECG, blood pressure, and arterial blood gases will be monitored continuously.

The video-guided PCT procedure requires extubation and re-intubation with the TVTTM tube.

Re-intubation with the TVTTM tube will be performed as any commonly practiced intubation.

The ETView Tracheoscopic system (TVTTM) consists of an ETT, embedded with a video imaging device and a light source at its tip and an integrated cable with a connector, that may be wired to any video monitor.

The imaging system will be used to monitor the airways while intubating and, beyond the vocal cords, to locate the transtracheal insertion site and needle. In addition, the light source will serve for transillumination of the neck soft tissues, in order to delineate the tracheal curvature and identify anatomical deviations.

Anesthesia and analgesia will be routinely performed, and standardized for all the study patients. Low doses of the opiate fentanyl (2-3 μg/kg) and the short-acting sedative propofol (20 mg bolus, and 3-6mg/kg/h drip) will be administered at the beginning of the procedure. Rocuronium bromide, a brief acting muscle paralyzer, 0.6mg/kg, will also be used in most patients.

Patient follow-up

The executing physician will answer a questionnaire evaluating the intraprocedural difficulties, complications, feasibility, confidence, and operability. A second physician, blinded to the procedure performed, will monitor the study patients during the first 6h after the procedure, or until discharge. Follow-up will include documentation of any procedure-related complications, monitoring of respiratory/ventilatory parameters and length of stay (LOS) in the ICU beyond 6h (due to medical circumstances related to the procedure).

All study patients will be placed with arterial lines through which we withdraw blood before and after the procedure, and when indicated by deterioration of respiratory parameters - for blood gas analyses (PaO2/FiO2, PaCO2, pH and BE). In addition, saturation will be documented hourly, and all patients will have chest x-rays performed immediately following tracheostomy.

Safety will be assessed by the frequency of procedure-related complications. These include:

A. Technical complications: False route/paratracheal insertion, injury to a thoracic vessel, tracheal/laryngeal/esophageal injury, accidental decannulation, puncturing the cuff, inserting the guide wire through Murphy's eye, malpositioning or kinking of the tracheal cannula, failed tracheostomy, multiple punctures (≥3).

B. Clinical complications potentially related to the procedure:

B.1. Intraprocedural: endotracheal bleeding (>100cc) and transfusion requirements (RBC, FFP or platelets), transient hypoxia/hypoxemia, hemodynamic changes (e.g., transient hypotension not related to anesthetics).

B.2. Postprocedure: alterations in respiratory function (defined as >15% reduction in saturation or PaO2/FiO2, compared to baseline; Increased PaCO2 without change in saturation; the need to change ventilatory settings and/or add PEEP within the first 24 hrs), atelectasis, pneumothorax, pneumomediastinum, aspiration, early unexplained mortality (within the first 24 hrs).

Operability will be evaluated via a questionnaire answered by the executing intensivist (enclosed within proposal documents). The main parameters they will be asked to evaluate will be: whether the transtracheal needle was recognized via the TVTTM (yes/no); intraoperative difficulties; number of technical complications; level of confidence; ease of performance ("best practice"); and need to convert to surgical tracheostomy procedure.

In addition, another member of the team will measure operative time, which includes the total duration of the procedure; the time it took to recognize the tracheal insertion site and needle; and the time to perform the PCT, that we define as the time since ETT placement until successful tracheal placement is confirmed via air bubbles or ETCO2.

Study size

A power analysis for time to perform the PCT as the primary endpoint, with 80% power to detect a 5 minute reduction in this outcome and significance of 0.05 or greater, indicates that at least 17 patients would be required in each group. We wish to enroll 30 patients for each group.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will enroll for this study
* patients aged >18 years old, admitted to the ICU,
* who require elective PCT for prolonged mechanical ventilation, airway protection or weaning failure.

Exclusion Criteria:

* Patients indicated for surgical tracheostomy, due to altered or difficult local anatomy;
* necessity of emergency airway access due to acute airway compromise;
* evidence of infection in the soft tissues of the neck;
* coagulation abnormalities (INR>1.5, PTT>40, thrombocyte count < 50,000);
* gross distortion of the neck anatomy (due to hematoma/tumor/thyromegaly/scarring from previous neck surgery/ unstable C-spine);
* contra-indication for re-intubation/suspected loss of airway during re-intubation; hemodynamic instability.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
procedure-related complications | 6h

SECONDARY OUTCOMES:
operative time | minutes

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sorkine, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Idit Matot, MD, Study Chair — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel